CLINICAL TRIAL: NCT04979884
Title: Safety and Therapeutic Efficacy of Cyclosporine Plus Standard of Care Treatment on ARDS in COVID -19 Patients at Alexandria University Hospitals in 2021: a Comparative Study
Brief Title: Safety and Effectiveness of Cyclosporin in the Management of COVID19 ARDS Patients in Alexandria University Hospital
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Science and Technology Development Fund (STDF), ,Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cyclosporine in COVID-19
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Cytokine Release Syndrome; Pulmonary Fibrosis
Keywords: COVID-19; Cyclosporine; secondary haemophagocytic lymphohistiocytosis (sHLH); acute respiratory distress syndrome (ARDS)
MeSH Terms: conditions — Cytokine Release Syndrome; Pulmonary Fibrosis; COVID-19; Respiratory Distress Syndrome | interventions — Cyclosporine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- cyclosporine (Experimental): patients will receive cyclosporine + (standard care treatment (± anticoagulant± antibiotic± antipyretic± steroid) according to Alexandria university hospitals protocol )
  Interventions: Drug: cyclosporine
- Standard of care treatment (Active Comparator): patients will receive standard treatment (antiviral ± anticoagulant± antibiotic± antipyretic± steroid± interleukin ) according to Alexandria university hospitals protocol.
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: cyclosporine — Dose of Cyclosporine oral capsule of 6 mg/kg/day divided into two doses with normal kidney function for 8-14 days
  Other Names: interleukin-2

SUMMARY:
The study to evaluate the effect of cyclosporine ( IL2 inhibitor and antiviral) verse standard care treatment on decrease ADRS, hyper inflammation, hypercytokinemia, and the mortality rate

DETAILED DESCRIPTION:
To test the efficacy of IL-2 inhibitors (Cyclosporine) compared to the Standard of care according to hospital protocol on COVID-19 patients concerning the clinical outcome (cytokines level, clinical improvement, and PCR of SARS-CoV-2 through the study period).

AIM:

The slow progression of the disease, improving survival among COVID-19 patients, and Standard assessment of patient improvement.

* Standard assessment of patient improvement:
* PCR-SARS-CoV-2 negative
* No fever
* No cytopenia (Hb ≥90 g/L, ANC ≥0.5x109/L, platelets ≥100x109/L) •
* No hyperferritinemia ≥500 μg/L
* (Decrease of IL2)

ELIGIBILITY:
Inclusion Criteria:

1. Current infection with COVID-19
2. written informed consent
3. Confirmed diagnosis of COVID-19 by PCR (polymerase chain reaction) tests and/or Positive Serology or any existing and validated diagnostic COVID-19 parameters during this time.
4. 18yrs ≥ Age <66 yrs
5. Chest X-ray showing suggestive of COVID-19 disease.
6. Both gender
7. The presence of Pulmonary fibrosis or hyper inflammation signs or A syndrome of cytokine release defined as any of the following::

   1. Leukopenia or lymphopenia,
   2. Ferritin > 500ng/mL or D-dimers ≥ 500 ng/mL
   3. Hs>90

Exclusion Criteria:

1. Lactation and Pregnancy women
2. unlikely to survive beyond 48h
3. Need for mechanical ventilation.
4. cases of multiorgan failure or abnormal renal function and shock.
5. malignancies, autoimmune disease, Perforation of the bowels or diverticulitis.
6. active bacterial or fungal infection.
7. We define impairment of cardiac function as poorly controlled heart diseases, cardiac insufficiency, unstable angina pectoris, myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia needs treatment or intervention, Uncontrolled hypertension (>180/110 mmHg.
8. Levels of serum transaminase >5 upper references rang
9. Symptoms of active tuberculosis or human immunodeficiency virus (HIV) positivity
10. the patient receiving Vaccines: Live, attenuated vaccines
11. Subjects received monoclonal antibodies within one week before admission.
12. Patients receiving high-dose systemic steroids (> 20 mg methylprednisolone or equivalent), immunosuppressant or immunomodulatory drugs
13. Contraindications for use in people with psoriasis include concomitant treatment with methotrexate, other immunosuppressant agents, coal tar, or radiation therapy.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with a 6-point ordinal scale showing each severity level | 7-14 days after randomization
  i. Death ii. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation iii. Hospitalized, on non-invasive ventilation or high flow oxygen devices iv. Hospitalized, requiring supplemental oxygen v. Hospitalized, not requiring supplemental oxygen vi. Not hospitalized

SECONDARY OUTCOMES:
Duration of hospital admission | through study completion, an average of 4 weeks
  efficacy of CsA (cyclosporine) in reducing days in hospital
Rate of decline OF Soluble interleukin-2 (IL-2) receptor alpha. (sCD25) | Days 1, 8, 15 or at hospital discharge(through study completion, an average of 6 weeks)
  change from baseline in IL-2 levels
Rate of decline OF interleukin-1 | Days 1, 8, 15 or at hospital discharge(through study completion, an average of 6 weeks)
  change from baseline in IL-1 levels
Rate of decline OF interleukin-10(IL-10) | Days 1, 8, 15 or at hospital discharge(through study completion, an average of 4 weeks)
  change from baseline in IL-10 levels
Rate of decline OF Interleukin-6,( IL-6) | Days 1, 8, 15 or at hospital discharge(through study completion, an average of 4 weeks)
  change from baseline in IL-6levels
Rate of decline OF Tumour necrosis factor α (TNFα) | Days 1, 8, 15 or at hospital discharge(through study completion, an average of 4 weeks)
  change from baseline in TNFα levels
Time to 50% a decrease of ferritin levels compared to peak value during trial | up to 28 days
  change from baseline in ferritin levels
Lung imaging improvement time | up to 28 days
  COVID19 Lung imaging determination
Time for non-invasive or invasive initial use | during hospital admission (up to 28 days)]
  efficacy of CSA in reducing days of ventilators
Time to improvement in oxygenation | up to 28 days) from hospitalization
  defined as independence from supplemental oxygen
Number of days safe from ventilators | during hospital admission (up to 28 days)
  efficacy of CSA in reducing days of ventilators
Number of days on mechanical ventilation | during hospital admission (up to 28 days)
  to evaluate the efficacy of CSA in reducing days of ventilators
Number of days in the intensive care unit after randomization | during hospital admission (up to 28 days)]
  to evaluate the efficacy of CSA in reducing days in the intensive care unit
Incidence of (Adverse Events) and Incidence of nosocomial bacterial or invasive fungal infection | during hospital admission (up to 28 days)]
  to evaluate the safety of CSA
Mean change of SOFA score in ICU patients | between 1, 15 days) hospital discharge
  The Sequential Organ Failure Assessment (SOFA) score: 0 (best) - 24 (worse) The SOFA score will be used to assess the probability of organ failure and mortality in ICU patients
Mean improvement in Clinical Deterioration Changed Early Warning Score (MEWS) between 1, 15 days) | between 1, 15 days) hospital discharge
  efficacy of CsA in Clinical improvement
rate of Mortality | throughout 30 and 90 days
  efficacy of CsA in reducing mortality
all-cause mortality will be measured. | At 28, 30, and 90 days,
  efficacy of CsA in reducing mortality

CONTACTS AND LOCATIONS:
Overall Officials: Maged El-Setouhy, Study Director — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fellman CL, Archer TM, Wills RW, Mackin AJ. Effects of cyclosporine and dexamethasone on canine T cell expression of interleukin-2 and interferon-gamma. Vet Immunol Immunopathol. 2019 Oct;216:109892. doi: 10.1016/j.vetimm.2019.109892. Epub 2019 Jul 11. PMID 31446206
- [Background] Damaso CR, Keller SJ. Cyclosporin A inhibits vaccinia virus replication in vitro. Arch Virol. 1994;134(3-4):303-19. doi: 10.1007/BF01310569. PMID 8129618
- [Background] Ciesek S, Steinmann E, Wedemeyer H, Manns MP, Neyts J, Tautz N, Madan V, Bartenschlager R, von Hahn T, Pietschmann T. Cyclosporine A inhibits hepatitis C virus nonstructural protein 2 through cyclophilin A. Hepatology. 2009 Nov;50(5):1638-45. doi: 10.1002/hep.23281. PMID 19821520